CLINICAL TRIAL: NCT03274076
Title: Evaluation of Tofacitinib in Early Diffuse Cutaneous Systemic Sclerosis (dcSSc): A Phase I/II Two Center Safety and Tolerability Study
Brief Title: Evaluation of Tofacitinib in Early Diffuse Cutaneous Systemic Sclerosis (dcSSc)
Acronym: TOFA-SSc
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Dinesh Khanna, MD, MS, Frederick G L Huetwell Professor of Rheumatology and Professor of Internal Medicine, Medical School, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00131837
Record Dates: First submitted 2017-08-28; First posted 2017-09-06 (Actual); Results first posted 2020-05-08 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-04

CONDITIONS: Systemic Sclerosis; Scleroderma
Keywords: diffuse; scleroderma; systemic sclerosis
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse | interventions — tofacitinib

STUDY DESIGN:
Intervention Model Description: Eligible subjects will be randomized to tofacitinib or placebo in a 2:1 manner.
Who Masked: Participant, Investigator
Masking Description: The study staff (with the exception of the study pharmacist) and the patient are blinded to the treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tofacitinib (Active Comparator): 5mg Tofacitinib twice a day
  Interventions: Drug: Tofacitinib
- Placebo (Placebo Comparator): 5mg Placebo twice a day
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Tofacitinib — Oral medication tofacitinib 5 mg twice a day for 24 weeks.
  Other Names: Xeljanz
  Arms: Tofacitinib
Drug: Placebo Oral Tablet — Oral Placebo 5 mg twice a day for 24 weeks
  Arms: Placebo

SUMMARY:
This Phase I/II placebo controlled trial will evaluate tofacitinib in subjects with diffuse cutaneous systemic scleroderma (dcSSc). This trial is intended to provide safety, and tolerability data in participants with dcSSc when dosed to target exposures similar to that used in adult participants with rheumatoid arthritis.

DETAILED DESCRIPTION:
The purpose of this clinical research study is to evaluate the safety, tolerability and efficacy of treatment with tofacitinib (study drug) versus placebo (a substance with no active ingredients and therefore may have no treatment benefit) in people with diffuse cutaneous systemic scleroderma. Subjects will be randomized to tofacitinib vs. placebo in a 2:1 ratio at 5 mg twice a day for 24 weeks. Subjects will then be offered to participate in an open label phase during which they will receive tofacitinib 5 mg twice a day for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of systemic sclerosis (SSc), as classified using the 2013 American College of Rheumatology/ European Union League Against Rheumatism classification of SSc.
2. Diffuse Cutaneous Systemic Sclerosis (dcSSc) as defined by 2001 LeRoy and Medsger
3. Disease duration ≤ 60 months (defined as time from the first non-Raynaud phenomenon manifestation)
4. Modified Rodnan Skin Score (mRSS) units ≥ 10 and ≤ 45 at screening.
5. Agreement to receive varicella-zoster vaccination (Zostavax®) or have received vaccination prior to screening.
6. Oral corticosteroids (≤ 10 mg/day of prednisone or equivalent) are permitted if the patient is on a stable dose regimen for ≥ 2 weeks prior to and including the baseline visit.
7. Ability to provide informed consent.

Exclusion Criteria:

1. Rheumatic disease other than dcSSc; it is acceptable to include patients with fibromyalgia, Sjogren syndrome, and scleroderma-associated myopathy
2. Limited cutaneous SSc or sine scleroderma
3. Major surgery (including joint surgery) within 8 weeks prior to baseline.
4. Any infected ulcer at screening
5. Subjects with any serious bacterial infection within the last 3 months, unless treated and resolved with antibiotics, or any chronic bacterial infection (e.g., chronic pyelonephritis, osteomyelitis, or bronchiectasis)
6. Oral corticosteroids >10 mg/day of prednisone or equivalent.
7. Hydroxychloroquine >400 mg/day, methotrexate >25 mg/week, D-Penicillamine >1000mg/day or mycophenolate mofetil > 2 grams/day prior to baseline. **Subjects can be on combination therapy of hydroxychloroquine and methotrexate or hydroxychloroquine and mycophenolate mofetil and must have been on a stable dose for at least 1 month prior to baseline visit.
8. Prior history of treatment in the 3 months prior to baseline with biological disease modifying anti-rheumatic drugs (DMARDs)potent immunosuppressants such as cyclosporine and azathioprine
9. Treatment with etanercept within ≤ 2 weeks of baseline: infliximab, certolizumab, golimumab, abatacept, tocilizumab, or adalimumab within ≤ 8 weeks of baseline; and anakinra within ≤ 1 week prior to the baseline visit.
10. Intravenous corticosteroids within 2 weeks prior to baseline visit.
11. Treatment with any investigational agent ≤ 4 weeks prior to baseline (or 5 half-lives of the investigational drug, whichever is longer)
12. Other investigational or marketed biologics with immunomodulatory properties within 3 months prior to baseline.
13. Treatment with anti-CD20 6 months prior to baseline and B cell counts <LLN
14. Any prior treatment with cell-depleting therapies other than anti-CD20 such as CAMPATH, anti-CD4, anti-CD5, anti-CD3, anti-CD19
15. Any prior treatment with chlorambucil, bone marrow transplantation, or total lymphoid irradiation
16. Vaccinated or exposed to a live/attenuated vaccine (other than Zostavax®) ≤ 6 weeks prior to baseline; or is expected to be vaccinated or to have household exposure to these vaccines during treatment or during the 6 weeks following discontinuation of study medication. (**See additional inclusion for obtaining Zostavax® prior to entering the study)
17. Pulmonary disease with Forced Vital Capacity (FVC) ≤ 50% of predicted, or Diffusing capacity of the lungs for carbon monoxide (DLCO),(uncorrected for hemoglobin) ≤ 40% of predicted
18. History of pulmonary arterial hypertension (PAH) with mean PAP> 30 mmHg on right heart catheterization requiring subcutaneous or intravenous prostacyclin or dual use of oral PAH therapies
19. Subjects at risk for tuberculosis (TB):

    A. Specifically excluded from this study will be participants with a history of active TB within the last 3 years, even if it was treated; a history of active TB greater than 3 years ago, unless there is documentation that the prior anti-TB treatment was appropriate in duration and type; current clinical, radiographic, or laboratory evidence of active TB; (TB results within 30 days of screening will be accepted and will not to be repeated. B. Latent TB at or within 30 days of screening, history of or current positive purified protein derivative tuberculin skin test (PPD) ( >5mm induration, regardless of Bacille Calmette Guerin [BCG] vaccine and/or QuantiFERON Gold, a negative chest x-ray, and no symptoms or risk factors), unless one month of prophylaxis has been completed prior to inclusion
    * An indeterminate QuantiFERON® unless followed by a subsequent negative PPD or negative QuantiFERON® or a consultation with and clearance by local infectious disease (ID) department is required.
20. Positive for hepatitis B surface antigen at or within 30 days of screening
21. Positive for hepatitis C antigen at or within 30 days of screening
22. Current or recent history of uncontrolled clinically significant renal, hepatic, hematologic, gastrointestinal, metabolic, endocrine, pulmonary, cardiac or neurologic disease.
23. History of human immunodeficiency virus (HIV), (as determined by medical records or patient reported).
24. History of diverticulitis or chronic, ulcerative lower gastrointestinal (GI) disease such as Crohns disease, ulcerative colitis, or other symptomatic, lower GI conditions that might predispose a patient to perforations.
25. Pregnant or breastfeeding female subjects; and female subjects of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in the protocol for the duration of the study and for at least 28 days after discontinuation of study drug.
26. Severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase risk associated with study participation and in the judgment of the investigator would make the subject inappropriate for entry into this study.
27. History of systemic sclerosis (SSc) Renal Crisis within the 6 months prior to baseline.
28. Any of the following lab results at screening:

    * Hemoglobin <9 g/dL or Hematocrit <30%
    * White Blood Cell count <3.0 x 109/L;
    * Absolute Neutrophil count <1.2 x 109/L;
    * White Blood Cell count <3.0 x 109/L;
    * Absolute Neutrophil count <1.2 x 109/L;
    * Platelet count <100 x 109/L;
    * Absolute Lymphocyte count <0.75 x 109/L.
    * ALT or AST > 1.5 × the upper limit of normal (ULN) of normal at screening or any uncontrolled clinically significant laboratory abnormality that would affect interpretation of study data or the patient's participation in the study
    * Total bilirubin > upper limit of normal (ULN) at Screening.
    * Estimated glomerular filtration rate [GFR] <40mL/min/1.73 m2
29. Prior rituximab use without documentation of normalized b cell counts.
30. History of recurrent (more than one episode) herpes zoster or disseminated (at least one episode) herpes zoster, or disseminated (at least one episode) herpes simplex
31. History of any lymphoproliferative disorder, such as Epstein Barr Virus (EBV) related lymphoproliferative disorder, history of lymphoma, leukemia, or signs and symptoms suggestive of current lymphatic disease.
32. History of any malignancy in the last 5 years with the exception of adequately treated or excised basal cell or squamous cell or cervical cancer in situ.
33. Significant trauma or surgery procedure within 1 month prior to first dose of study drug.
34. History of alcohol or substance abuse, unless in full remission for greater than 6 months prior to first dose of study drug.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh Khanna, MD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Khanna D, Padilla C, Tsoi LC, Nagaraja V, Khanna PP, Tabib T, Kahlenberg JM, Young A, Huang S, Gudjonsson JE, Fox DA, Lafyatis R. Tofacitinib blocks IFN-regulated biomarker genes in skin fibroblasts and keratinocytes in a systemic sclerosis trial. JCI Insight. 2022 Sep 8;7(17):e159566. doi: 10.1172/jci.insight.159566. PMID 35943798

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from University of Michigan and University of Pittsburgh Scleroderma clinics. The recruitment period began in September 2017 and ended with the last participant randomization in October 2018.
Groups:
- Tofacitinib Double Blind 0-24 Weeks: Participants treated with an oral medication tofacitinib 5 mg twice daily for 24 weeks with option to enter 24 weeks of open label tofacitinib.
- Placebo Double Blind 0-24 Weeks: Participants treated with an oral placebo 5 mg twice daily for 24 weeks with option to enter 24 weeks of open label tofacitinib.
- Tofacitinib to Tofacitinib Open Label 24-48 Weeks; Placebo to Tofacitinib Open Label 24-48 Weeks: Post double blind completion, participants receive 5mg tofacitinib twice daily for 24 weeks.
Period: 24 Weeks Double Blind
Arm/Group | Tofacitinib Double Blind 0-24 Weeks | Placebo Double Blind 0-24 Weeks | Tofacitinib to Tofacitinib Open Label 24-48 Weeks | Placebo to Tofacitinib Open Label 24-48 Weeks
Started | 10 | 5 | 0 | 0
Completed | 10 | 4 | 0 | 0
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Period: 24 Weeks Open Label
Arm/Group | Tofacitinib Double Blind 0-24 Weeks | Placebo Double Blind 0-24 Weeks | Tofacitinib to Tofacitinib Open Label 24-48 Weeks | Placebo to Tofacitinib Open Label 24-48 Weeks
Started | 0 | 0 | 10 | 4
Completed | 0 | 0 | 8 | 3
Not Completed | 0 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo Double Blind 0-24 Weeks: Participants treated with oral placebo tablet 5 mg twice a daily for 24 weeks with option to enter 24 weeks of open label tofacitinib.
- Total: Total of all reporting groups
Arm/Group | Tofacitinib Double Blind 0-24 Weeks | Placebo Double Blind 0-24 Weeks | Total
Number analyzed (Participants) | 10 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (13.9) | 60.0 (9.7) | 50.8 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 5 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 10 | 4 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Study was conducted only in the United States
  Participants
    United States | 10 | 5 | 15
Disease Duration [Mean (Standard Deviation); unit: years] | 2.0 (1.3) | 2.4 (1.2) | 2.1 (1.2)
Baseline Modified Rodnan Skin Score (mRSS [Mean (Standard Deviation); unit: units on a scale] — The Modified Rodnan Skin Score (mRSS) is a measure of skin thickness. Skin thickness in 17 anatomic areas was rated on a 0-3 scale and scores are summed to obtain the mRSS (range from 0 - 51), with higher mRSS scores indicating worse skin involvement.
  units on a scale | 22.7 (9.3) | 24.4 (6.9) | 23.3 (8.4)
Forced Vital Capacity (FVC) % Predicted [Mean (Standard Deviation); unit: percent predicted] — Forced Vital Capacity (FVC) is the amount of air that can be forcibly exhaled after a full breath and is a measure of lung function. Predicted FVC was based on institutional standards. Values lower than 80% are indicated as abnormal.
  percent predicted | 90.7 (16.5) | 83.8 (17.5) | 88.4 (16.6)
Diffusion in liters of carbon monoxide (DLCO) % Predict [Mean (Standard Deviation); unit: percent predicted] — Diffusion in liters of carbon monoxide (DLCO) is a measure of lung function. Predicted values for DLCO were computed using the Crapo Morris equations. Values lower than 80% are considered abnormal.
  percent predicted | 82.4 (19.7) | 92.0 (20.5) | 85.6 (19.8)
Health Assessment Questionnaire - Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: units on a scale] — Health Assessment Questionnaire - Disability Index (HAQ-DI) is a self-reported questionnaire of functionality that includes questions in 8 domains (dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities). The final score ranges from 0 to 3, where a higher HAQ-DI score indicates a worse outcome.
  units on a scale | 1.01 (0.6) | 0.80 (0.5) | 0.98 (.59)
Proportion of Participants with Tender Friction Rubs [Count of Participants; unit: Participants] — Tender Friction Rubs are noticeable upon exam and show as grating sensations to the fibrinous deposits on the surface of the tendon sheaths and overlying fascia
  Participants | 1 | 1 | 2
Proportion of Participants with Large Joint Contractures [Count of Participants; unit: Participants] — Large joint contracture is caused by shortening of muscles, tendons, ligaments, and joint capsules or by heterotopic ossification that affect the large joints.
  Participants | 5 | 0 | 5
Proportion of Participants with Background Immunosuppressive [Count of Participants; unit: Participants] — Background medications included within the immunosuppressive group included: methotrexate and mycophenolic acid.
  Participants | 9 | 4 | 13
Proportion of Participants Using Prednisone [Count of Participants; unit: Participants] | 2 | 2 | 4
Proportion of Participants with Interstitial Lung Disease on High-resolution computed tomography [Count of Participants; unit: Participants] — High-resolution computed tomography (HRCT) is a type of computed tomography with specific techniques to enhance image resolution. It is used in the diagnosis of various health problems, though most commonly for diseases of the lung.
  Participants | 4 | 2 | 6
Proportion of Participants with Small Joint Contractures [Count of Participants; unit: Participants] — Small joint contracture is caused by shortening of muscles, tendons, ligaments, and joint capsules or by heterotopic ossification that affect the small joints.
  Participants | 9 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience Grade 3 or Higher Adverse Events That Occur at or Before Week 24
Description: Primary outcome is met if any participants experience a grade 3 or higher event prior to Week 24. A grade 3 AE would constitute as "severe". Grading was following using CTCAE v 4.03.
  Note that the planned statistical analysis (Fisher's exact test) could not be performed because there were no events.
Time Frame: 24 weeks
Population: All participants were included in this analysis although 1 placebo participant withdrew prior to week 24. They remained in the intent to treat population.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Double Blind 0-24 Weeks: Participants treated with oral placebo tablet 5 mg twice a day for 24 weeks with option to enter 24 weeks of open label tofacitinib.
Arm/Group | Tofacitinib Double Blind 0-24 Weeks | Placebo Double Blind 0-24 Weeks
Number analyzed (Participants) | 10 | 5
Participants | 0 | 0

2. Secondary Outcome: Number of Grade 3 (Severe) or Higher Adverse Events That Occur Throughout the Study
Description: Grade 3 or higher adverse events (AEs) assessed throughout the study ( 48 weeks). A grade 3 AE would constitute as "severe". Grading was following using CTCAE v 4.03.
  Note that the planned statistical analysis (calculation of rate ratio and 90% CI) could not be performed at Weeks 12 and 24 due to no events, and could not be performed at Week 36 because there were no events in the placebo group (denominator).
Time Frame: Week 12, 24, 36, and 48
Population: One placebo participant withdrew prior to week 24. 1 additional placebo participant and 2 tofacitinib participants withdrew prior to week 48 but after completing week 24 and entering the open label portion.
Measure: Number; unit: Adverse Events
Groups:
- Tofacitinib Double Blind 0-24 Weeks: Participants treated with an oral medication tofacitinib 5mg twice daily for 24 weeks with option to enter 24 weeks of open label tofacitinib.
- Placebo Double Blind 0-24 Weeks: Participants treated with an oral placebo tablet 5mg twice daily for 24 weeks with option to enter 24 weeks of open label tofacitinib.
Arm/Group | Tofacitinib Double Blind 0-24 Weeks | Placebo Double Blind 0-24 Weeks | Tofacitinib to Tofacitinib Open Label 24-48 Weeks | Placebo to Tofacitinib Open Label 24-48 Weeks
Number analyzed (Participants) | 10 | 5 | 10 | 4
Adverse Events
  Week 12: number analyzed (Participants) | 10 | 5 | 0 | 0
  Week 12 | 0 | 0 |  |
  Week 24: number analyzed (Participants) | 10 | 4 | 0 | 0
  Week 24 | 0 | 0 |  |
  Week 36: number analyzed (Participants) | 0 | 0 | 8 | 3
  Week 36 |  |  | 2 | 0
  Week 48: number analyzed (Participants) | 0 | 0 | 8 | 3
  Week 48 |  |  | 1 | 1
Statistical Analysis 1: Comparison: Tofacitinib to Tofacitinib Open Label 24-48 Weeks vs Placebo to Tofacitinib Open Label 24-48 Weeks; H0: Rate of grade 3 (severe) or higher adverse events that occur throughout week 48 in Placebo = Rate of grade 3 (severe) or higher adverse events that occur throughout week 48 in Tofacitinib; Test type: Superiority; Rate ratio = 1.25, 90% CI 2-sided [0.19 to 8.33] — Tofacitinib represents the numerator, and placebo represents the denominator

3. Secondary Outcome: Number of Grade 2 (Moderate) or Higher Adverse Events That Occur Throughout the Study
Description: Grade 2 or higher assessed 12 weeks apart. Grade 2 AEs are determined as " moderate". Grading was performed following CTCAE v 4.03 guidance.
Time Frame: Week: 12, 24, 36, and 48
Population: One placebo participant withdrew prior to week 24. 1 additional placebo participant and 2 tofacitinib participants withdrew prior to week 48 but after completing week 24.
Measure: Number; unit: Adverse Events
Groups:
- Tofacitinib to Tofacitinib Open Label 24-48 Weeks; Placebo to Tofacitinib Open Label 24-48 Weeks: Post double blind completion, participants receive 5 mg tofacitinib twice daily for 24 weeks.
Arm/Group | Tofacitinib Double Blind 0-24 Weeks | Placebo Double Blind 0-24 Weeks | Tofacitinib to Tofacitinib Open Label 24-48 Weeks | Placebo to Tofacitinib Open Label 24-48 Weeks
Number analyzed (Participants) | 10 | 5 | 10 | 4
Adverse Events
  Week 12: number analyzed (Participants) | 10 | 5 | 0 | 0
  Week 12 | 7 | 5 |  |
  Week 24: number analyzed (Participants) | 10 | 4 | 0 | 0
  Week 24 | 5 | 5 |  |
  Week 36: number analyzed (Participants) | 0 | 0 | 8 | 3
  Week 36 |  |  | 14 | 3
  Week 48: number analyzed (Participants) | 0 | 0 | 8 | 3
  Week 48 |  |  | 4 | 1
Statistical Analysis 1: Comparison: Tofacitinib Double Blind 0-24 Weeks vs Placebo Double Blind 0-24 Weeks; H0: Rate of grade 2 (moderate) or higher adverse events that occur throughout week 12 in Placebo = Rate of grade 2 (moderate) or higher adverse events that occur throughout week 12 in Tofacitinib; Test type: Superiority; Rate ratio = 0.65, 90% CI 2-sided [0.25 to 1.71] — Tofacitinib represents the numerator, and Placebo represents the denominator
Statistical Analysis 2: Comparison: Tofacitinib Double Blind 0-24 Weeks vs Placebo Double Blind 0-24 Weeks; H0: Rate of grade 2 (moderate) or higher adverse events that occur throughout week 24 in Placebo = Rate of grade 2 (moderate) or higher adverse events that occur throughout week 24 in Tofacitinib; Test type: Superiority; Rate ratio = 0.53, 90% CI 2-sided [0.26 to 1.07] — Tofacitinib represents the numerator, and Placebo represents the denominator
Statistical Analysis 3: Comparison: Tofacitinib to Tofacitinib Open Label 24-48 Weeks vs Placebo to Tofacitinib Open Label 24-48 Weeks; H0: Rate of grade 2 (moderate) or higher adverse events that occur throughout week 36 in Placebo = Rate of grade 2 (moderate) or higher adverse events that occur throughout week 36 in Tofacitinib; Test type: Superiority; Rate ratio = 0.85, 90% CI 2-sided [0.49 to 1.49] — Tofacitinib represents the numerator, and Placebo represents the denominator
Statistical Analysis 4: Comparison: Tofacitinib to Tofacitinib Open Label 24-48 Weeks vs Placebo to Tofacitinib Open Label 24-48 Weeks; H0: Rate of grade 2 (moderate) or higher adverse events that occur throughout week 48 in Placebo = Rate of grade 2 (moderate) or higher adverse events that occur throughout week 48 in Tofacitinib; Test type: Superiority; Rate ratio = 0.89, 90% CI 2-sided [0.52 to 1.52] — Tofacitinib represents the numerator, and Placebo represents the denominator

4. Secondary Outcome: Number of Adverse Events of Special Interest (AESI) Throughout the Study
Description: AESI are pre-defined adverse events as indicated in the protocol. They include: infections, stomach perforations, malignancy, herpes zoster and lab abnormalities.
  Note that the planned statistical analysis (calculation of rate ratio and 90% CI) could not be performed at Weeks 12 and 24 because there were no events in placebo group (denominator).
Time Frame: Weeks 12, 24, 36 and 48
Population: Placebo participant withdrew prior to week 24. 1 additional placebo participant and 2 tofacitinib participants withdrew prior to week 48.
Measure: Number; unit: Adverse Events
Groups:
- Tofacitinib Double Blind 0 - 24 Weeks: Participants treated with an oral medication tofacitinib 5mg twice daily for 24 weeks with option to enter 24 weeks of open label tofacitinib.
- Placebo Double Blind 0 - 24 Weeks: Participants treated with an oral placebo tablet 5mg twice daily for 24 weeks with option to enter 24 weeks of open label tofacitinib.
Arm/Group | Tofacitinib Double Blind 0 - 24 Weeks | Placebo Double Blind 0 - 24 Weeks | Tofacitinib to Tofacitinib Open Label 24-48 Weeks | Placebo to Tofacitinib Open Label 24-48 Weeks
Number analyzed (Participants) | 10 | 5 | 10 | 4
Adverse Events
  Week 12: number analyzed (Participants) | 10 | 5 | 0 | 0
  Week 12 | 4 | 0 |  |
  Week 24: number analyzed (Participants) | 10 | 5 | 0 | 0
  Week 24 | 1 | 0 |  |
  Week 36: number analyzed (Participants) | 0 | 0 | 8 | 3
  Week 36 |  |  | 4 | 1
  Week 48: number analyzed (Participants) | 0 | 0 | 8 | 3
  Week 48 |  |  | 0 | 1
Statistical Analysis 1: Comparison: Tofacitinib to Tofacitinib Open Label 24-48 Weeks vs Placebo to Tofacitinib Open Label 24-48 Weeks; H0: Rate of adverse events of special interest throughout week 36 in Placebo = Rate of adverse events of special interest throughout week 36 in Tofacitinib; Test type: Superiority; Rate ratio = 3.85, 90% CI 2-sided [0.68 to 21.77] — Tofacitinib represents the numerator, and Placebo represents the denominator
Statistical Analysis 2: Comparison: Tofacitinib to Tofacitinib Open Label 24-48 Weeks vs Placebo to Tofacitinib Open Label 24-48 Weeks; H0: Rate of adverse events of special interest throughout week 48 in Placebo = Rate of adverse events of special interest throughout week 48 in Tofacitinib; Test type: Superiority; Rate ratio = 1.87, 90% CI 2-sided [0.5169 to 6.7652] — Tofacitinib represents the numerator, and Placebo represents the denominator

5. Secondary Outcome: Change in Modified Rodnan Skin Score (mRSS)
Description: The Modified Rodnan Skin Score (mRSS) is a measure of skin thickness. Skin thickness in 17 anatomic areas was rated on a 0-3 scale and scores are summed to obtain the mRSS (range from 0 - 51), with higher mRSS scores indicating worse disease activity
Time Frame: Change from Baseline at weeks: 12, 24, 36, and 48
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Tofacitinib Double Blind 0-24 Weeks: .Participants treated with an oral medication tofacitinib 5mg twice daily for 24 weeks with option to enter 24 weeks of open label tofacitinib.
- Tofacitinib (DB Tofacitinib) Open Label 24 - 48 Weeks; Tofacitinib (DB Placebo) Open Label 24-48 Weeks: Post double blind completion, participants receive 5mg tofacitinib twice daily for 24 weeks.
Arm/Group | Tofacitinib Double Blind 0-24 Weeks | Placebo Double Blind 0-24 Weeks | Tofacitinib (DB Tofacitinib) Open Label 24 - 48 Weeks | Tofacitinib (DB Placebo) Open Label 24-48 Weeks
Number analyzed (Participants) | 10 | 5 | 8 | 3
score on a scale
  Week 12: number analyzed (Participants) | 10 | 5 | 0 | 0
  Week 12 | -2 [-4 to -1] | 0.5 [-2 to 4.5] |  |
  Week 24: number analyzed (Participants) | 10 | 5 | 0 | 0
  Week 24 | -5.5 [-6 to -1] | -2.5 [-7.5 to 2.5] |  |
  Week 36: number analyzed (Participants) | 0 | 0 | 8 | 3
  Week 36 |  |  | -10 [-12 to -4] | -6 [-9.5 to -2.5]
  Week 48: number analyzed (Participants) | 0 | 0 | 8 | 3
  Week 48 |  |  | -12.5 [-15.5 to -5.5] | -9 [-11 to -9]
Statistical Analysis 1: Comparison: Tofacitinib Double Blind 0-24 Weeks vs Placebo Double Blind 0-24 Weeks; H0: The absolute change in mRSS from week 0 to week 12 in placebo = The absolute change in mRSS from week 0 to week 12 in Tofacitinib; Test type: Superiority; p = 0.1978, Exact Wilcoxon
Statistical Analysis 2: Comparison: Tofacitinib Double Blind 0-24 Weeks vs Placebo Double Blind 0-24 Weeks; H0: The absolute change in mRSS from week 0 to week 24 in placebo = The absolute change in mRSS from week 0 to week 24 in Tofacitinib; Test type: Superiority; p = 0.4665, Exact Wilcoxon
Statistical Analysis 3: Comparison: Tofacitinib (DB Tofacitinib) Open Label 24 - 48 Weeks vs Tofacitinib (DB Placebo) Open Label 24-48 Weeks; H0: The absolute change in mRSS from week 0 to week 36 in placebo = The absolute change in mRSS from week 0 to week 36 in Tofacitinib; Test type: Superiority; p = 0.3063, Exact Wilcoxon
Statistical Analysis 4: Comparison: Tofacitinib (DB Tofacitinib) Open Label 24 - 48 Weeks vs Tofacitinib (DB Placebo) Open Label 24-48 Weeks; H0: The absolute change in mRSS from week 0 to week 48 in placebo = The absolute change in mRSS from week 0 to week 48 in Tofacitinib; Test type: Superiority; p = 0.6000, Exact Wilcoxon

6. Secondary Outcome: Provisional American College of Rheumatology Combined Response Index (CRISS) Systemic Sclerosis
Description: CRISS components included the following domains: modified Rodnan skin score, forced vital capacity percent predicted, Physician Global Assessment, Patient Global Assessment, and Health Assessment Questionnaire Disability-Index. An algorithm determines the predicted probability of improvement from baseline by incorporating change in the mRSS, FVC percent predicted, Physician and Patient Global Assessments, and HAQ-DI. The outcome is a continuous variable between 0.0 and 1.0 (0 - 100%). A cut-off at 0.6 in the predicted probability of being improved has yielded the smallest misclassification error. Subjects are not considered improved if, between Visit 1 and 6, they develop new: 1) renal crisis; 2) decline in FVC% predicted by 15% (relative) from baseline and confirmed after 1 month; or 3) left ventricular failure (systolic ejection fraction < 45%) or pulmonary artery hypertension. Higher CRISS scores indicates improvement.
Time Frame: Week:12, 24, and 48
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Tofacitinib Double Blind 0-24 Weeks | Placebo Double Blind 0-24 Weeks | Tofacitinib to Tofacitinib Open Label 24-48 Weeks | Placebo to Tofacitinib Open Label 24-48 Weeks
Number analyzed (Participants) | 10 | 5 | 10 | 4
score on a scale
  Week 12: number analyzed (Participants) | 10 | 5 | 0 | 0
  Week 12 | 0.07 [0.005 to 0.35] | 0.02 [0.001 to 0.28] |  |
  Week 24: number analyzed (Participants) | 10 | 5 | 0 | 0
  Week 24 | 0.28 [0.001 to 1.00] | 0.09 [0.02 to 0.56] |  |
  Week 48: number analyzed (Participants) | 0 | 0 | 10 | 4
  Week 48 |  |  | 0.99 [0.33 to 1.00] | 0.83 [0.53 to 1.00]
Statistical Analysis 1: Comparison: Tofacitinib Double Blind 0-24 Weeks vs Placebo Double Blind 0-24 Weeks; H0: The CRISS score at week 12 in placebo = The CRISS score at week 12 in Tofacitinib; Test type: Superiority; p = 0.4535, Exact Wilcoxon
Statistical Analysis 2: Comparison: Tofacitinib Double Blind 0-24 Weeks vs Placebo Double Blind 0-24 Weeks; H0: The CRISS score at week 24 in placebo = The CRISS score at week 24 in Tofacitinib; Test type: Superiority; p = 0.8392, Exact Wilcoxon
Statistical Analysis 3: Comparison: Tofacitinib to Tofacitinib Open Label 24-48 Weeks vs Placebo to Tofacitinib Open Label 24-48 Weeks; H0: The CRISS score at week 48 in placebo = The CRISS score at week 48 in Tofacitinib; Test type: Superiority; p = 0.9212, Exact Wilcoxon

ADVERSE EVENTS:
Time Frame: This report includes the entire time frame of the study with both Double Blind and Open Label = 48 weeks.
Description: Coding of adverse events into body system was performed by the study chair for adverse events and by the medical monitors for serious adverse events.
Arm/Group | Tofacitinib Double Blind 0-24 Weeks | Placebo Double Blind 0-24 Weeks | Tofacitinib to Tofacitinib Open Label 24-48 Weeks | Placebo to Tofacitinib Open Label 24-48 Weeks
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5 | 0/10 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5 | 3/10 | 1/4
Other Adverse Events (participants affected / at risk) | 9/10 | 5/5 | 9/10 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tofacitinib Double Blind 0-24 Weeks (N=10) | Placebo Double Blind 0-24 Weeks (N=5) | Tofacitinib to Tofacitinib Open Label 24-48 Weeks (N=10) | Placebo to Tofacitinib Open Label 24-48 Weeks (N=4)
Diabetic foot ulcer (non-infection), complicated by thermal injury. (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bells's Palsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus-induced Hepatitis, Drug-Induced Hepatitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Worsening SSc-Inpatient (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tofacitinib Double Blind 0-24 Weeks (N=10) | Placebo Double Blind 0-24 Weeks (N=5) | Tofacitinib to Tofacitinib Open Label 24-48 Weeks (N=10) | Placebo to Tofacitinib Open Label 24-48 Weeks (N=4)
Hypercholesterolemia (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Weight Gain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic Kidney Disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased GERD (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Otis Externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Digital Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ulcer Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bilateral Wrist Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Low Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive Urgency (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flu-like Symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-obstructive Renal Calculi (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
> 50% LDL/HDL (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Colititis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Left Hip Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intentional Weight Loss (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left Knee Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Right trochanteric bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle Weakness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpatations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Premature Ventricular Contractions (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Elevated Creatine Phosphokinase (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridemia (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug-induced hepatitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug Induced Hepatitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Worsening ILD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/76/NCT03274076/SAP_001.pdf
  • Study Protocol (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/76/NCT03274076/Prot_002.pdf